CLINICAL TRIAL: NCT03282110
Title: Comprehensive Acupuncture for Depressive Disorder With Comorbid Psychogenic Pain: Randomized Controlled Study
Brief Title: Comprehensive Acupuncture for Depressive Disorder With Comorbid Psychogenic Pain
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: China Academy of Chinese Medical Sciences (Other)
Responsible Party: Principal Investigator, Peijing Rong, The deputy director of Institute of Acupuncture and Moxibustion, China Academy of Chinese Medical Sciences, China Academy of Chinese Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ChinaACMS-3
Record Dates: First submitted 2017-08-28; First posted 2017-09-13 (Actual); Last update posted 2017-11-07 (Actual); Status verified 2017-09

CONDITIONS: Depression; Psychoneurotic; Pain
MeSH Terms: conditions — Depression; Pain | interventions — Citalopram

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ta-VNS & Electro-acupuncture (Experimental): 1. Device:ta-VNS(transcutaneous vagus nerve stimulation):2 times per day,5 consecutive days per week for two months
  2. Other:Electro-acupuncture:3 times per week, once every other day for two months
  Interventions: Device: ta-VNS; Other: Electro-acupuncture
- Citalopram (Active Comparator): citalopram for oral administration; 10mg for the first 1-3 days, 20mg for the following 4-7 days；40mg for the left days within two months
  Interventions: Drug: Citalopram

INTERVENTIONS:
Device: ta-VNS — The transcutaneous vagus nerve stimulation (taVNS) at auricular concha is a typical representative of TCM modernization. The taVNS regulates the autonomic nervous system, which shows a good therapeutic effect for the treatment of depression.
  Other Names: transcutaneous vagus nerve stimulation
  Arms: ta-VNS & Electro-acupuncture
Other: Electro-acupuncture — one of the most common acupuncture methods, selecting acupoints based on traditional Chinese medicine theory. It exerts the function to regulate qi and blood circulation and balance Yang and Yin energy inside body.
  Arms: ta-VNS & Electro-acupuncture
Drug: Citalopram — Citalopram is an antidepressant drug of the selective serotonin reuptake inhibitor (SSRI) class.It has U.S. Food and Drug Administration approval to treat major depression.
  Other Names: brand name：Cipramil, SFDA J20130028
  Arms: Citalopram

SUMMARY:
Experimental and clinical studies have indicated that acupuncture has a good effect for depression and comorbid pain. The purpose of this research is to compare the effect of comprehensive electro-acupuncture therapy and western medicine citalopram for for depressive disorder with comorbid psychogenic pain. This research is a assessor blinded, randomized controlled trials. 60 patients will be randomly divided into comprehensive electro-acupuncture group and western medicine citalopram for 8 weeks treatment and the therapeutic effect is done at the end of 1,2,4,6,8 week.

ELIGIBILITY:
Inclusion Criteria:

* Conform with the diagnostic criteria of depression according to DIAGNOSTIC AND STATISTICAL MANUAL OF MENTAL DISORDERS (DSM-5TM)
* Age from 18 to 50 year-old
* Patients with the first onset depression
* Patients with mild-to-moderate depression scored 12-30 by Montgomery scale
* Patients with one psychogenic pain at least, and the degree of VAS is 3 or more
* Volunteer participants willing to cooperate and obeying the treatment

Exclusion Criteria:

* Pregnant woman
* Patients with severe primary diseases and acute diseases of heart, brain, liver, kidney and hematopoietic systems and infectious disease, malignant tumor
* Patients who can't stop taking drugs according to the requirement in the treatment period
* Patients with a history of schizophrenia and other mental disorders
* Patients with cognitive impairment or personality disorders
* Patients have serious suicide idea or suicidal behavior

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-11-30 (Estimated); Primary Completion 2018-06-30 (Estimated); Study Completion 2019-06-30 (Estimated)

PRIMARY OUTCOMES:
Montgomery-Asberg Depression Rating Scale Change | Baseline and 1 week,baseline and 2 weeks,baseline and 4 weeks,baseline and 6 weeks,baseline and 8 weeks
  Measure the severity of depressive episodes in patients with mood disorders, It contents ten items, and each item is scored 0-6.(0=no depression,6=depression as bad as can be), yielding a total between 0 and 60.

SECONDARY OUTCOMES:
SF-McGill Pain Questionnaire | Baseline and 1 week,baseline and 2 weeks,baseline and 4 weeks,baseline and 6 weeks,baseline and 8 weeks
  Measure pain in 3 ways:1)pain rating indexes: pain intensity from feeling and emotional aspects, it includes fifteen items and each item is scored 0-3(0=no pain 3=severe) 2)present pain intensity, scored 0-5(0=no pain, 5=intense pain) 3)VAS: visual analog scale
SF-36 Health Survey Questionnaire | Baseline and 4 weeks, baseline and 8 weeks
  Measure the self-reported living quality.It has eight sections:the physiological function, physiological function, the body pain, general health, energy, social function, emotional function and mental health.It consists of eight scaled scores, which are the weighted sums of the questions in their section.
Pittsburgh Sleep Quality Index | Baseline and 1 week,baseline and 2 weeks,baseline and 4 weeks,baseline and 6 weeks,baseline and 8 weeks
  A self-report questionnaire that assesses sleep quality over a 1-month time interval. The measure consists of 19 individual items, creating seven components that produce one global score
Hamilton Anxiety Rating Scale(HAMA) | Baseline and 1 week,baseline and 2 weeks,baseline and 4 weeks,baseline and 6 weeks,baseline and 8 weeks
  A psychological questionnaire used by clinicians to rate the severity of a patient's anxiety.Each of the 14 items contains some symptoms, and each group of symptoms is rated on a scale of zero to four, with four being the most severe.

OTHER OUTCOMES:
Salivary cortisol levels | baseline and 8 weeks
  Serum cortisol levels positively correlated with the severity of depression, so that the saliva should be collected before and after treatment. Acquisition time of saliva: 7：30～8：30 am and 3:00-4:00 p.m
Physiological indexes | baseline and 8 weeks
  Including blood pressure, ECG, respiration, pulse check, blood routine, blood biochemistry, urine analysis to see if there is any change during treatment
Adverse events that are related to treatment | baseline and 8 weeks
  Measure the incidence of adverse events of acupuncture such as fainting during acupuncture treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Peijing Rong, Dotor, Study Director — Institute of Acupuncture and Moxibustion, China Academy of Chinese Medical Sciences; Zhangjing Zhang, Dotor, Study Director — The School of Chinese Medicine, The University of Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided